CLINICAL TRIAL: NCT06039488
Title: The Impact of an 8-week Exercise Program on Physical Function in Individuals With Cancer
Brief Title: Effectiveness of a Cancer Exercise Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Ciaran Fairman, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109975
Record Dates: First submitted 2023-09-05; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): 2 days/week of resistance and cardiovascular exercise for 8-weeks
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — A combination of resistance exercise and cardiovascular exercise (performed 2 days per week for 8-weeks) is tailored to each individual in accordance with their medical/cancer-related history, baseline assessments of physical function, and overall goals.
  Resistance exercise includes 6-8 exercises targeting major muscle groups. The first week of the program is used to familiarize participants to the exercises of the program, provide coaching on safe and appropriate technique, and identifying initial load for 2 sets of 12 repetitions (equivalent to ~65% 1 repetition maximum), with a goal of working towards 4 sets of 8 reps. Additionally, participants are asked to perform 20-30 minutes of moderate-to-vigorous aerobic activity (approximately 60-85% age-predicted heart rate maximum) via walking, jogging, or cycling each session.

SUMMARY:
The investigators are examining the impact of an 8-week multi-modal exercise program (resistance and cardiovascular training) delivered 2 times per week on physical function adults (>18 years old) with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 diagnosed with cancer

Exclusion Criteria:

* unwilling to come to the on-site clinic for exercise sessions
* any neuromuscular, cardiovascular, or psychological condition precluding safe exercise
* unable to read/understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Bellarmine Norton Assessment Tool (2-minute Step Test) | 0 and 8-weeks
  2-minute Step Test: Number of times an individuals' knee reaches a predetermined heigh during a 2-minute period of marching
Bellarmine Norton Assessment Tool (Timed Arm Curl) | 0 and 8-weeks
  Timed Arm Curl: Number of repetitions an arm curl individuals can complete in 30 seconds)
Bellarmine Norton Assessment Tool (30 second Chair Stand) | 0 and 8-weeks
  Chair Stand: Number of times participants can stand from a sitting position and return to sitting in 30 seconds

SECONDARY OUTCOMES:
Fatigue | 0 and 8-weeks
  The Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale: The FACIT-Fatigue scale is a 13-item scale that will be used to assess cancer-related fatigue. The FACIT-Fatigue scale is scored on a 0-4 response scale from 0 = "not at all" to 4 "very much", regarding items related to fatigue and energy in the past 7 days. Lower score indicates greater fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fairman CM, Harrington SE, Schumpp AR, Brooks AM, Jones MJ, Kim J, Kennedy MA. Planning and evaluating an integrated clinical exercise oncology service: an exploratory mixed-methods study. BMC Health Serv Res. 2024 Oct 31;24(1):1318. doi: 10.1186/s12913-024-11797-0. PMID 39478564